CLINICAL TRIAL: NCT00367055
Title: Comparison of the Action of the Rosiglitazone-metformin Fixed-dose Combination and of a Metformin-sulfonylurea Free Combination on the B-cell Function in Type 2 Diabetic Patients Not Controlled With Metformin Alone.
Brief Title: Rosiglitazone-Metformin Combination Versus Metformin-Sulfonylurea Combination On Beta-Cell Function In Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101765; AVAF4001
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Results first posted 2009-11-05 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Beta cell function; Type 2 diabetes; Combination treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination; Metformin

INTERVENTIONS:
Drug: rosiglitazone-metformin
Drug: Metformin
Drug: metformin+ gliclazide
  Other Names: rosiglitazone-metformin; Metformin

SUMMARY:
It has been shown in previous study that progressive glycemic deterioration was associated with progressive loss of b-cell function, measured by the decrease in plasma insulin levels, irrespective of the therapy used (diet, sulfonylureas or metformin).There is growing evidence that thiazolidinediones could have a positive action on the b-cell function. But it has not yet been demonstrated that they could protect from a deterioration in insulin secretion in the long term. So, it appears interesting to study the long term evolution of the b-cell function and the possible protection with rosiglitazone in patients with type 2 diabetes showing evidence of loss of b-cell function with metformin alone.

ELIGIBILITY:
INCLUSION CRITERIA:

* Males and females 40 to 75 years of age (inclusive at the time of screening)
* Type 2 diabetes mellitus as defined by the WHO criteria, diagnosed for at least 1 year
* Subjects receiving 1.5 to 3g of metformin alone at a constant dose for at least 8 weeks prior to visit 1
* Patients with 6.5% < HbA1c > 8% at visit 1 and visit 2
* 25 < BMI < 35

EXCLUSION CRITERIA:

* Patient with type 1 diabetes
* Treatment with other hypoglycaemic agents than metformin in the last 3 months
* FPG >200 mg/dL at visit 2
* Hypersensitivity to the studied treatments (rosiglitazone, metformin chlorhydrate, gliclazide)
* Congestive heart failure (NYHA class I to IV), unstable or severe angina, recent myocardial infarction
* Respiratory insufficiency
* Subjects who have required the use of insulin for glycaemic control in the past 6 months prior to visit 1 (except during pregnancy or acute episodes such as hospitalization, trauma or infection) or subjects with a history of metabolic acidosis including diabetic ketoacidosis
* Anemia defined by haemoglobin concentration <11.0 g/dL for males and <10.0 g/dL for females
* Renal disease or renal dysfunction, e.g. as suggested by serum creatinine levels ≥135.0 µmol/L in males and ≥110.0 µmol/L in females and/or creatinine clearance <40 mL/min
* Presence of clinically significant hepatic disease, with ALT, AST, total bilirubin, alkaline phosphatase >2.5 times the upper limit of the normal reference range
* Subjects with chronic diseases requiring periodic ot intermittent treatment with oral or IV corticosteroids
* Subjects receiving danazol, miconazole or phenylbutazone
* Active alcohol, drug or medication abuse within the last 6 months or any condition that would indicate the likelihood of poor subject compliance
* Women who are lactating, pregnant or planning to become pregnant
* Any clinically significant abnormality identified at screening which, in the investigator's judgement, makes the subject unsuitable for inclusion in the study
* Use of any other investigational agent within 30 days or 5 half-lives (whichever is longer) prior to visit 1
* Subjects who receive or anticipate receiving radiocontrast dye during the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosiglitazone + Metformin 4 mg/2 g/Day: Initial dose of rosiglitazone + metformin of 4 milligrams (mg)/2 grams (g)/day; allowed adjustment of up to 8 mg/2 g/day after 8 weeks
- Gliclazide + Metformin 80 mg/2 g/Day: Initial dose of gliclazide + metformin 80 mg/2 g/day; allowed adjustment of up to 160 mg/2 g/day after 4 weeks, up to 240 mg/2 g/day after 8 weeks, up to 320 mg/2 g/day after 3 months
Period: Overall Study
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Started | 43 | 41
Completed | 32 | 30
Not Completed | 11 | 11
Not completed — Adverse Event | 6 | 3
Not completed — Patient's Willing | 3 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Stopping Criterion Met | 0 | 1
Not completed — Participant Living too Far from Hospital | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day | Total
Number analyzed (Participants) | 43 | 41 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.4) | 58.1 (8.0) | 58.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 32 | 25 | 57
Body Mass Index (BMI) [Number; unit: kilograms per square meter (kg/m2)] — Number of participants with the indicated class of BMI at randomization
  kilograms per square meter (kg/m2)
    <25 | 3 | 0 | 3
    25-30 | 21 | 20 | 41
    >30 | 19 | 21 | 40
FBG [Mean (Standard Deviation); unit: Millimoles/Liter (mmol/L)] — Mean fasting blood glucose (FBG) levels were measured by blood draw
  Millimoles/Liter (mmol/L) | 9.10 (1.72) | 8.28 (1.11) | 8.70 (1.50)
HbA1c [Mean (Standard Deviation); unit: percentage] — Mean hemoglobin A1c (HbA1c) levels were measured by blood draw
  percentage | 7.5 (0.55) | 7.3 (0.55) | 7.4 (0.57)

OUTCOME MEASURES:

1. Primary Outcome: Median Change From Baseline in the Insulin Secretory Capacity After a 36-month Treatment
Description: Change from baseline in the insulin secretory capacity was measured by the assesment of blood insulin concentrations (conc.) using the hyperglycaemic clamp (HC) technique, per intravenous glucose perfusion by a catheter. Change from baseline for insulin conc peaks (highest conc level) was calculated as the Month 36 value minus the baseline value. Insulin secretion was assessed by calculating AUC during the first 10 minutes of HC (incremental and total AUC0-10 min) and the AUC after the first 10 minutes of the HC (10-180min).
Time Frame: Baseline and Month 36
Population: Intent-to-Treat (ITT) Population: participants receiving at least one dose of study drug with an available efficacy evaluation (HC at M18 or M36). The measurement was conducted on participants who had baseline and M18 and M36 HC test data available. Each HC was validated at both Baseline and Month 36, resulting in different "n"s for each category.
Measure: Median (Full Range); unit: picomoles/L per minute (pmol/L*min)
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Number analyzed (Participants) | 27 | 29
picomoles/L per minute (pmol/L*min)
  Total AUC(0-10 min), n=24, 26 | -3.9 [-688.3 to 2211.2] | -75.3 [-919.9 to 1507.1]
  Incremental AUC(0-10 min), n=22, 23 | 7.0 [-308.3 to 2781.2] | 74.6 [-822.2 to 1193.8]
  Total concentration peak(0-10 min), n=25, 26 | -8.6 [-89.6 to 386.5] | 3.6 [-121.2 to 52.3]
  Incremental concentration peak(0-10 min), n=24, 26 | -1.8 [-60.9 to 443.8] | 10.8 [-128.3 to 56.6]
  Total AUC(10-180 min), n=20, 24 | 40.6 [-411.9 to 500.2] | -21.2 [-344.2 to 787.3]
  Incremental AUC(10-180 min), n=19, 24 | 67.0 [-304.2 to 518.4] | 13.6 [-264.9 to 793.4]
  Total concentration peak(10-180 min), n=27, 29 | 7.9 [-223.0 to 286.1] | -9.3 [-120.5 to 229.4]
  Incremental concentation peak(10-180 min), n=25,29 | 10.8 [-232.3 to 198.6] | 11.5 [-116.9 to 231.6]
Statistical Analysis 1: Comparison: Rosiglitazone + Metformin 4 mg/2 g/Day vs Gliclazide + Metformin 80 mg/2 g/Day; Test type: Superiority or Other; p = 0.376, Van Elteren — p value is for Total AUC(0-10 min)
Statistical Analysis 2: Comparison: Rosiglitazone + Metformin 4 mg/2 g/Day vs Gliclazide + Metformin 80 mg/2 g/Day; Test type: Superiority or Other; p = 0.990, Van Elteren — p value is for Incremental AUC(0-10 min)

2. Secondary Outcome: Median Change From Baseline in the Ratio M/I After a 36-month Treatment
Time Frame: Baseline and Month 36
Reporting Status: Not Posted

3. Secondary Outcome: Median Change From Baseline in the Insulin Secretion Capacity After an 18-month Treatment
Description: Change from baseline was calculated as the Month 18 value minus the baseline value. Insulin secretion capacity is measured in blood (blood level of insulin) and is a response of the pancreatic beta-cells to hyperglycemia induced by a glucose IV bolus, then infusion. Hyperglycemic clamp (HC) is a reference technique to evaluate the initial and the secondary phases of insulin secretion.
Time Frame: Baseline and Month 18
Population: as for outcome 1
Measure: Median (Full Range); unit: pmol/L*min
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Number analyzed (Participants) | 30 | 31
pmol/L*min
  HC, Total AUC(0-10min), n=30, 31 | 18.3 [-1044.7 to 2211.2] | -32.3 [-919.9 to 1612.5]
  HC, Incremental AUC(0-10min), n=27, 26 | 22.3 [-308.3 to 2781.2] | 60.7 [-822.2 to 1193.8]
  HC, Total AUC(10-180min), n=26, 30 | 55.9 [-411.9 to 500.2] | -7.6 [-344.2 to 787.3]
  HC, Incremental AUC(10-180min), n=26, 29 | 72.9 [-304.2 to 518.4] | 14.6 [-264.9 to 1172.7]
  Arginine (Arg) test, Total AUC(0-30min), n=25, 25 | 38.4 [-367.0 to 225.0] | 10.9 [-163.9 to 93.1]
  Arg test, Incremental AUC(0-30min), n=25, 25 | 15.1 [-440.3 to 120.9] | -8.0 [-153.3 to 49.3]
  Arg test, Incremental Conc. peak(0-30 min),n=26,29 | 23.3 [-2531.7 to 766.5] | -111.1 [-1125.0 to 499.7]

4. Secondary Outcome: Mean Change From Baseline in HbA1c at Month 36
Description: Change from baseline was calculated as the Month 36 value minus the baseline value. HbA1c levels were measured by blood draw.
Time Frame: Baseline and Month 36
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug and had an available efficacy evaluation (hyperglycaemic clamp at M18 or M36). This measurement was conducted on participants in the ITT Population who had baseline and M18 and M36 clamp test data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Number analyzed (Participants) | 32 | 31
percent change | -0.22 (1.3) | 0.3 (1.2)

5. Secondary Outcome: Mean Change From Baseline in FBG at Month 36
Description: Change from baseline was calculated as the Month 36 value minus the baseline value. FBG levels were measured by blood draw.
Time Frame: Baseline and Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Number analyzed (Participants) | 32 | 30
millimoles per Liter (mmol/L) | -1.6 (1.9) | -0.2 (2.4)

6. Secondary Outcome: Median Change From Baseline in Insulin Resistance Index (HOMA-IR) After a 36-month Treatment
Time Frame: Baseline and Month 36
Reporting Status: Not Posted

7. Secondary Outcome: Median Change From Baseline in Beta Cell Function Index (HOMA-beta) After a 36-month Treatment
Time Frame: Baseline and Month 36
Reporting Status: Not Posted

8. Secondary Outcome: Mean Change From Baseline in CPP Total and Incremental AUC T0-T30 After a 36-month Treatment
Time Frame: Baseline and Month 36
Reporting Status: Not Posted

9. Secondary Outcome: Mean Change From Baseline in CPP Concentration Peak and Incremental Concentration Peak T0-T30 After a 36-month Treatment
Time Frame: Baseline and Month 36
Reporting Status: Not Posted

10. Secondary Outcome: Mean Change From Baseline in Insulin Sensitivity Index at Months 18 and 36
Description: Change from baseline was calculated as the Month 18 and 36 values minus the baseline value. Insulin sensitivity is measured as the quantity of glucose metabolized per unit of plasma insulin concentration.
Time Frame: Baseline and Months 18 and 36
Population: ITT Population
Measure: Mean (Standard Deviation); unit: micromoles (umol)/kilogram/min/pmol/L
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Number analyzed (Participants) | 30 | 33
micromoles (umol)/kilogram/min/pmol/L
  Month 18 | -0.00511 (0.03451) | -0.02045 (0.05302)
  Month 36 | 0.00040 (0.04722) | -0.01702 (0.05109)

ADVERSE EVENTS:
Arm/Group | Rosiglitazone + Metformin 4 mg/2 g/Day | Gliclazide + Metformin 80 mg/2 g/Day
Serious Adverse Events (participants affected / at risk) | 8/43 | 12/41
Other Adverse Events (participants affected / at risk) | 31/43 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone + Metformin 4 mg/2 g/Day (N=43) | Gliclazide + Metformin 80 mg/2 g/Day (N=41)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute on chronic (Gastrointestinal disorders) | 1 | 0
Partial bowel obstruction (Gastrointestinal disorders) | 0 | 1
Proctorrhagia (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Urinary incontinence aggravated (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Digital necrosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Myocardial ischemia (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Peritoneal carcinomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone + Metformin 4 mg/2 g/Day (N=43) | Gliclazide + Metformin 80 mg/2 g/Day (N=41)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Common cold (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lumbago (Musculoskeletal and connective tissue disorders) | 4 | 1
Lumbar pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Gonalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 4
Carpal tunnel syndrome (Nervous system disorders) | 1 | 4
Sciatica (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 1
Formication (Nervous system disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 1
Sigmoiditis (Gastrointestinal disorders) | 2 | 1
Colopathy (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Tonsilitis (Infections and infestations) | 1 | 2
Fungal infection (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 0 | 3
Orchitis (Infections and infestations) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.